CLINICAL TRIAL: NCT03314298
Title: A Single Dose Trial to Evaluate the Pharmacokinetics of Testosterone and Anastrozole From Subcutaneous Testosterone and Anastrozole (T+Ai) in Premenopausal Women
Brief Title: A Single Dose Trial to Evaluate the Pharmacokinetics of Testosterone and Anastrozole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Havah Therapeutics Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HAV-001
Record Dates: First submitted 2017-08-06; First posted 2017-10-19 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2017-10

CONDITIONS: Mammographic Density
MeSH Terms: interventions — Testosterone; Anastrozole

STUDY DESIGN:
Intervention Model Description: open labelled pharmacokinetic study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- testosterone anastrozole implant (Experimental): testosterone 80mg Anastrozole 4 mg single as a subcutaneous pellet
  Interventions: Drug: testosterone anastrozole

INTERVENTIONS:
Drug: testosterone anastrozole — subcutaneous testosterone and anastrozole
  Other Names: testosterone; anastrozole

SUMMARY:
A single dose trial to evaluate the pharmacokinetics of testosterone and anastrozole from subcutaneous testosterone and anastrozole (T+Ai) in premenopausal women

DETAILED DESCRIPTION:
The trial is of open label single centre design. The serum concentrations of testosterone and plasma concentrations of anastrozole will be measured in 12 premenopausal women. Participants will be stratified in a 50:50 manner in two BMI (Body Mass Index) groups, <25 and 25 kg/m2, respectively. There will be a lead group of two participants in whom the serum/plasma concentrations will be examined after the first four weeks, to determine whether the sampling schedule adequately describes the serum/plasma concentration-time profiles or should be adjusted.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to and be capable of understanding and signing an Informed Consent Form.
2. Patients seeking treatment with Investigational Product for the reduction in high mammographic breast density (MBD).
3. Pre-menopausal levels of Follicular stimulating hormone/Leutinizing hormone/estradiol(follicle stimulating hormone/luteinizing hormone/oestrogen) according to the definition of "pre-menopausal range" for the laboratory involved.
4. Volpara Density volumetric breast density of ≥15.5% (combined average both breasts)
5. Age between 35-55 years inclusive.
6. Body weight between 50-90 kg inclusive.
7. BMI between 20-30 kg/m2 inclusive.
8. Good venous access for venepuncture.
9. In good general health without clinically significant cardiac, respiratory, or psychiatric disease.
10. Negative pregnancy test in women of childbearing potential (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilisation), no more than seven days before the first dose of Investigational Product.
11. For women of childbearing potential who are sexually active, agreement to use a highly effective, non-hormonal form of contraception (Mirena (TM) allowed) during and for at least six months after completion of treatment with Investigational Product; OR, a fertile male partner willing and able to use effective non-hormonal means of contraception (barrier method of contraception in conjunction with spermicidal jelly, or surgical sterilisation) during and for at least six months after completed dosing Investigational Product.

Exclusion Criteria:

1. Presence of breast cancer.
2. Previous or concomitant other malignancy (non-breast, other than skin) within the previous five years.
3. Diabetes mellitus or glucose intolerance defined as a fasting glucose of ≥ 6 mmol/L.
4. History of coronary artery disease.
5. Risk of transmitting Human Immunodeficiency Virus or viral hepatitis via infected blood.
6. Existing testosterone, oestrogen and/or anastrozole treatment.
7. Concomitant medication which induces or inhibits CYP3A4 (Listed in Appendix A).
8. Current warfarin usage.
9. Prolonged systemic corticosteroid treatment, inhalation and topical steroids allowed.
10. Known hypersensitivity to any component of Investigational Product.
11. Systemic reproductive hormone replacement therapy.
12. Systemic hormonal contraception.
13. Participation in another clinical trial of an Investigational Product within 30 days of entry into the present trial or within 4-5 half-lives of the Investigational Product, whichever is the longer.
14. Use of any product containing ginseng within 30 days of screening.
15. Pregnant or lactating women.
16. Unable to comply with trial requirements.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
testosterone Cmax | Day 1, blood samples will be taken pre-dose and at 1, 2, 4, 8 and 12 hours and 9 am in the morning on Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57, 71 and 85.
  Peak Plasma Concentration
testosterone AUC | Day 1, blood samples will be taken pre-dose and at 1, 2, 4, 8 and 12 hours and 9 am in the morning on Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57, 71 and 85.
  Area under the plasma concentration versus time curve
testosterone T1/2 | Day 1, blood samples will be taken pre-dose and at 1, 2, 4, 8 and 12 hours and 9 am in the morning on Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57, 71 and 85.
  plasma half-life
anastrozole Cmax | Day 1, blood samples will be taken pre-dose and at 1, 2, 4, 8 and 12 hours and 9 am in the morning on Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57, 71 and 85.
  Peak Plasma Concentration
anastrozole AUC | Day 1, blood samples will be taken pre-dose and at 1, 2, 4, 8 and 12 hours and 9 am in the morning on Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57, 71 and 85.
  Area under the plasma concentration versus time curve
anastrozole T1/2 | Day 1, blood samples will be taken pre-dose and at 1, 2, 4, 8 and 12 hours and 9 am in the morning on Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57, 71 and 85.
  plasma half-life

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | The outcome measures will be reported weekly until study completion-3 months
  To assess the safety and tolerability of T+Ai following a single dose of T+Ai by subcutaneous implantation.
  Biochemical and hematological will be evaluated and the number of participants with abnormal values or adverse events that are related to treatment will be recorded
dihydrotestosterone metabolism | 3 months
  To description of the time course of dihydrotestosterone serum concentrations.
breast elasticity | Breast tissue elasticity will be measured by shear wave ultrasound at baseline and on Days 29, 57 and 85
  Breast tissue elasticity will be measured by shear wave ultrasound at baseline and on Days 29, 57 and 85. A Supersonic Ultrasound will be carried out by four quadrant analysis of each breast with 6x3mm Q box analyses measured in kPa.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Birrell, Md PhD, Principal Investigator — Wellend Health
Locations (1):
- Wellend Health, Toorak Gardens, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided